CLINICAL TRIAL: NCT00739635
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Evaluation of the Efficacy, Safety and Tolerability of Neramexane in Patients With Subjective Tinnitus
Brief Title: Efficacy, Safety and Tolerability of Neramexane in Patients With Subjective Tinnitus
Acronym: EASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ 92579/TI/3001; EudraCT Number 2007-007835-16
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Subjective Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Neramexane mesylate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neramexane mesylate — Double-blind treatment period of 17 weeks up to 75 mg Neramexane mesylate per day
  Arms: 1
Drug: Placebo — Double-blind treatment period of 17 weeks placebo
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of neramexane mesylate in the treatment of subjective tinnitus in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years with a clinical diagnosis of first onset,
* Persistent (i.e. tinnitus should never be absent for > 24 hours in a row), subjective, uni- or bilateral tinnitus present for at least 3 months but not more than 12 months

Exclusion Criteria:

* Clinical diagnosis of intermittent or pulsatile tinnitus
* Patients who have tinnitus as a concomitant symptom of an otological/neurological disease (such as otitis media, Menière's disease, otosclerosis, etc)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
TBF-12 (Tinnitus-Beeinträchtigungs-Fragebogen-12 "Tinnitus Handicap Inventory-12") total score change from baseline to end of treatment | Screening, Baseline, week 5, 13, 17

SECONDARY OUTCOMES:
TBF-12 factorial scores, individual responder rate, Tinnitus Rating Scale, Sleep Questionnaire, population pharmacokinetics, optional pharmacogenetics | 17 weeks
safety parameters | 17 weeks

CONTACTS AND LOCATIONS:
Locations (54):
- Austria (5):
  - Krankenhaus der Elisabethinen, Graz
  - Bezirkskrankenhaus Kufstein, Kufstein
  - A. ö. Krankenhaus der Elisabethinen Linz, Linz
  - Salzburger Landeskrankenhaus, Universitätsklinik für Hals-Nasen-Ohren-Krankheiten, Salzburg
  - Clin Pharm International GmbH, Zentrum Wien, Vienna
- Germany (25):
  - Dr. Elisabeth Kühne, Halle, Saale
  - Dr. med. Nobert Pasch, Aachen
  - Dr. Peter Küppers, Augsburg
  - Charité, Universitätsmedizin Berlin-Tinnituszentrum, Berlin
  - Klin. Forschung Berlin Buch GmbH, Berlin
  - Dr. med. Frank Reintjes, Braunschweig
  - ClinPharm International, Chemnitz
  - Dr. Klaus Peter Jayme, Darmstadt
  - Dr. Christian Dörr, Dresden
  - HNO-Praxis im Gesundheitszentrum Walsum, Duisburg
  - ClinPharm International GmbH, Frankfurt
  - ClinPharm International GmbH, Görlitz
  - Dr. Werner Gieselmann, Heiligenhaus
  - Dr. Wolfgang Lotte, Iserlohn
  - ClinPharm International GmbH, Leipzig
  - HNO Praxis, Lichtenfels
  - Dr. Dannesberger, Lorsch
  - ClinPharm International, Magdeburg
  - HNO Gemeinschaftpraxis, Meppen
  - LMU München Klinik Großhadern, Munich
  - Dr. med. Ulrike Walter, Nuremberg
  - Dr. Susanne Wiedemann, Nuremberg
  - Dr. Norbert Staab, Schlüchtern
  - Dr. Hannelore Neumaier, Wiesbaden
  - Dr. med. Stephanie Göbel, Worms
- Portugal (2):
  - Hospital Militar Regional nº 1 Serviço de Otorrinolaringologia, Porto
  - Clínica ORL Dr. Eurico de Almeida, Porto
- Spain (12):
  - Clínica Universitaria de Navarra, Dept. ORL, Pamplona, Navarre
  - Hospital Sagunto, Sagunto, Valencia
  - Fundación Hospital de Alcorcón, Otorhinolaryngology, Alcorcón - Madrid
  - Hospital Clínico Barcelona, Dept. Of ORL, Barcelona
  - Clinica Clivina, Private Consultancy, Jaén
  - Hospital Comarcal San Agustin, Linares, Jaén
  - Hospital Xeral-Calde, Lugo
  - Hospital Puerta del Hierro, Madrid- Servicio de OR, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Hospital Universtiario Son Dureta, Palma de Mallorca
  - Hospital Universitario de Salamanca- Hospital Virgen de la Vega, Salamanca
  - Hospital Universitario Virgen del Rocio- Centro de Especialidades Dr. Fleming, Seville
- United Kingdom (10):
  - Oldfield Surgery, Bath
  - Avondale Surgery Research office, Chesterfield
  - The Horsley Medical Practice, East Horsley, Leatherhead, Surrey
  - The university Hospitals of Leicester, Leicester Royal Infirmary, Leicester
  - Burbage Surgery, Leicestershire
  - The Freeman Hospital, Newcastle upon Tyne
  - Wansford and Kings Cliffe Practice, Petereborough
  - Frome Medical Practice, Somerset
  - Dr. Trevor Gooding, Warwick Shire
  - Sherbourne Medical Centre, Warwickshire

REFERENCES:
- See also: Related Info — http://www.merz.com